CLINICAL TRIAL: NCT00006156
Title: FSH-Stimulated Inhibin B as a Marker for Early Ovarian Insufficiency
Brief Title: Feasibility Study for Development of an Early Test for Ovarian Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Principal Investigator, Lawrence Nelson, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 000189; 00-CH-0189
Record Dates: First submitted 2000-08-09; First posted 2000-08-10 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-03

CONDITIONS: Healthy; Premature Ovarian Failure
Keywords: Ovarian Failure; Ovary; Aging; Healthy Volunteer; Primary Ovarian Insufficiency(POI); Premature Menopause; Premature Ovarian Failure (POF)
MeSH Terms: conditions — Primary Ovarian Insufficiency; Menopause, Premature

ARMS (2):
- Control (Experimental): Control for FSH stimulation test
  Interventions: Other: Control
- Drug: FSH (Experimental): FSH Stimulation Test
  Interventions: Drug: Drug: FSH

INTERVENTIONS:
Other: Control — No injection of FSH
  Arms: Control
Drug: Drug: FSH — FSH Stimulation Test
  Arms: Drug: FSH

SUMMARY:
This purpose of this study is to gain information about normal ovarian function that will be useful in developing a test for early detection of ovarian failure. The ovaries produce female hormones, such as estrogen, that are important in maintaining a woman's health. When the ovaries do not work properly, problems can develop. Unfortunately, there is no test that can detect ovarian failure early in its course. By the time premature ovarian failure is diagnosed in young women, two-thirds have already developed osteopenia (loss of some bone mass) and nearly one in ten have osteoporosis, a greater loss of bone mineral density that weakens bones and increases the risk of fractures.

Women with normal ovarian function ages 18 to 55 and postmenopausal women 60 years of age or older may be eligible for this study. Candidates will be screened with a medical history, physical examination, blood tests and vaginal ultrasound examination. For the ultrasound study, a probe that emits sound waves is inserted into the vagina, and the sound waves are converted to form images of the ovaries. The procedure is done with an empty bladder and takes about 10 minutes. After this screening visit (Visit 1), those enrolled in the study will return to the NIH Clinical Center for the following additional procedures:

Visit 2-Will be scheduled between days 3 and 5 of the menstrual cycle (for women who are still menstruating). Participants will have blood tests to measure hormone levels and to check for pregnancy, and will have another transvaginal ultrasound examination. They will then receive an injection of a synthetic form of follicle stimulating hormone (FSH), a hormone the body makes normally.

Visits 3 and 4-Will be scheduled 24 and 36 hours after the FSH injection given during Visit 2 for collection of blood samples.

Visit 5-Will be scheduled 48 hours after the FSH injection for additional blood sampling and a final transvaginal ultrasound examination.

DETAILED DESCRIPTION:
This is a pilot project to test the feasibility of developing an FSH stimulation test. There is a need for a sensitive and specific marker to detect ovarian insufficiency early in its course. FSH stimulates inhibin B production by the granulosa cells of the cohort of ovarian follicles; serum inhibin B in turn participates in the negative feedback loop regulating FSH secretion. This protocol is characterizing the normal FSH-stimulated serum inhibin B response to a single subcutaneous injection of 300 IU human recombinant FSH given on day 2 to 4 of the menstrual cycle. In preliminary analysis under this protocol we have demonstrated that FSH-stimulated serum inhibin B levels measured at 24 hours after injection is a more robust marker of functional ovarian age than ovarian follicle count by transvaginal ultrasound, basal serum Mullerian Inhibiting Substance (MIS) levels, or basal serum FSH levels. Multiple regression analysis has revealed that FSH-stimulated inhibin B, FSH-stimulated estradiol, and basal FSH contribute significantly to an ability to predict functional ovarian age (as approximated by chronological age). The resulting regression equation relating these three parameters with age has a correlation coefficient of 0.742 and a coefficient of determination of 0.551. The protocol is now evaluating the reproducibility of this test and the feasibility of generating normative data in young women between the ages of 18 and 25. The results of this study may define parameters that could lead to earlier diagnosis and treatment of premature ovarian insufficiency.

ELIGIBILITY:
* INCLUSION CRITERIA:

A. Women with normal ovarian function:

Age 18 to 55.

Normal body mass index (18-30 kg/m(2)).

Normal menstrual cycles (between 25-35 days in length).

Ovulatory serum progesterone concentrations (in excess of 6 ng/mL in the menstrual cycle just preceding the study cycle).

B. Postmenopausal women (to serve as negative controls):

Greater than or equal to 60 years of age.

Proven fertility (as evidenced by a history of pregnancy regardless of outcome).

Normal body mass index (18-30 kg/m(2)).

Naturally menopausal: amenorrhea for at least one year; serum FSH greater than 40 IU/mL.

C. Women carriers of FMR1 premutations:

Age 18 to 40.

50 to 200 CGG repeats.

Normal menstrual cycles (between 25-35 days in length).

Have previously had genetic counseling regarding their FMR1 status.

EXCLUSION CRITERIA:

History of infertility or infertility in a first degree relative.

Acute or chronic disease.

Menopause due to surgery, radiation, or chemotherapy.

Current use of oral contraceptives or hormone replacement therapy, or use of these agents within the previous 3 months.

Use within the previous three months of any medication known to affect the hypothalamic-pituitary-ovarian axis (including over-the-counter and alternative medicines).

History of excessive exercise (greater than 10 hours a week).

Girls will be excluded because there are no data regarding FSH use in children.

Smokers.

Pregnant.

Breast feeding.

Persistent ovarian masses.

History of tumors of the ovary, breast, uterus, hypothalamus, or pituitary.

History of breast or endometrial cancer.

History of hypersensitivity to recombinant FSH or any one of its excipients.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2000-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anasti JN, Kalantaridou SN, Kimzey LM, Defensor RA, Nelson LM. Bone loss in young women with karyotypically normal spontaneous premature ovarian failure. Obstet Gynecol. 1998 Jan;91(1):12-5. doi: 10.1016/s0029-7844(97)00583-8. PMID 9464713
- [Background] Coulam CB, Adamson SC, Annegers JF. Incidence of premature ovarian failure. Obstet Gynecol. 1986 Apr;67(4):604-6. PMID 3960433
- [Background] Faddy MJ, Gosden RG. A model conforming the decline in follicle numbers to the age of menopause in women. Hum Reprod. 1996 Jul;11(7):1484-6. doi: 10.1093/oxfordjournals.humrep.a019422. PMID 8671489

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug - FSH | Control
Started | 42 | 7
Completed | 42 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug - FSH | Control | Total
Number analyzed (Participants) | 42 | 7 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 7 | 48
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 7 | 49
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 40 | 4 | 44
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 29 | 3 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Follicle Stimulating Hormone Stimulated Serum Inhibin B Levels.
Time Frame: 24 hours
Measure: Mean (Standard Error); unit: participants
Arm/Group | Drug - FSH | Control
Number analyzed (Participants) | 42 | 7
participants
  Baseline | 50.7 (3.7) | 48.8 (8.8)
  24 Hours | 96.6 (7.9) | 47.7 (10.7)

2. Secondary Outcome: Follicle Stimulating Hormone Stimulated Serum Estradiol (E2) Levels
Time Frame: 24 hours
Measure: Mean (Standard Error); unit: participants
Arm/Group | Drug - FSH | Control
Number analyzed (Participants) | 42 | 7
participants
  Baseline | 29.9 (2.0) | 25.0 (3.4)
  24 Hours | 70.8 (6.4) | 28.3 (6.1)

ADVERSE EVENTS:
Groups:
- Adverse Events Not Collected: Adverse Events Not Collected
Arm/Group | Adverse Events Not Collected
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No